CLINICAL TRIAL: NCT02183454
Title: Multinational Abluminal Sirolimus Coated BiO-Engineered StenT - The MASCOT Post Marketing Registry
Brief Title: MASCOT - Post Marketing Registry
Acronym: MASCOT
Status: Completed | Type: Observational
Sponsor: OrbusNeich (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: VP-0639
Record Dates: First submitted 2014-06-26; First posted 2014-07-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: intracoronary stent; drug eluting stent; sirolimus; endothelial progenitor cells
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: OrbusNeich COMBO stent — The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.

SUMMARY:
To collect post marketing surveillance data on patients receiving at least one Combo Bio-Engineered Sirolimus Eluting Stent when used according to the Instructions for Use. Data will be collected in order to assess the long term safety and performance of the Combo Stent in routine clinical practice.

DETAILED DESCRIPTION:
The multicenter, multinational, prospective registry population consists of patients who undergo percutaneous coronary intervention (PCI) with (attempted) placement of at least one Combo Stent (according to the Instructions for use) as part of routine clinical care. Approximately 2,500 patients from 50 centers in Europe and Asia will be entered into the registry. Patients entered into the registry are followed for one year. The registry is considered finished when all patients have completed the 12 month follow-up.

A follow-up is scheduled at 30 days, 6 months and 12 months post procedure. Follow-up is obtained at a planned regular visit to the outpatient clinic, or by telephone contact with the patient.

ELIGIBILITY:
In general, consecutive patients are included in the registry. Patients are only excluded from registration if ANY of the following conditions apply:

1. Undergoing PCI for treatment of stent thrombosis
2. High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
3. Currently participating in another investigational drug or device study in which a routine angiographic follow-up is planned
4. A life expectancy of <12 months
5. Explicit refusal of participation in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who undergo PCI with (attempted) placement of at least one Combo Stent as part of routine clinical care are entered into the registry. PCI with a Combo Stent is considered attempted when the operator has passed the Combo Stent across the guiding catheter.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Adjudicated device-oriented composite target lesion failure (TLF) | 12 months post procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a non-target vessel, or ischemia-driven target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting (CABG)) at 12 months post procedure.

SECONDARY OUTCOMES:
Adjudicated TLF | at index procedure, 30 days, 6 months and 12 months post procedure
Each of the components of TLF (Cardiac death, Non-fatal MI not clearly attributable to a non-target vessel, Target lesion revascularization (TLR)) | at index procedure, 30 days, 6 months, 12 months
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) as a composite of all Death, any MI and ischemia-driven revascularization (TLR/TVR/non-TVR) | at index procedure, 30 days, 6 months and 12 months
Each of the components of MACE (All death, Any myocardial infarction, Ischemia-driven revascularization) | at index procedure, 30 days, 6 months and 12 months
Adjudicated stent thrombosis per the Academic Research Consortium (ARC) definition | at index procedure, 30 days, 6 months and 12 months post-procedure
Adjudicated bleeding per the Bleeding Academic Research Consortium (BARC) definition | at index procedure, 30 days, 6 months and 12 months post-procedure
Adjudicated stroke | at index procedure, 30 days, 6 months and 12 months
Device success: Percentage of patients with a successful delivery and deployment of the Combo Stent to the target lesion and a final diameter stenosis after stenting ≤20% by visual assessment in the presence of grade 3 TIMI flow, by visual estimation | Index Procedure
Procedure success: Successful stent placement and no peri-procedural complications. | Index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — San Raffaele Hospital
Locations (1):
- Amphia Ziekenhuis, Breda, Netherlands

REFERENCES:
- [Derived] Chandrasekhar J, Sartori S, Aquino MB, Baber U, Hajek P, Atzev B, Hudec M, Ong TK, Mates M, Borisov B, Warda HM, den Heijer P, Wojcik J, Iniguez A, Coufal Z, Khashaba A, Schee A, Munawar M, Gerber RT, Yan BP, Tejedor P, Kala P, Liew HB, Lee M, Kalkman DN, Dangas GD, de Winter RJ, Colombo A, Mehran R; MASCOT investigators (Appendix I). Comparison of One-Year Outcomes in Patients >75 Versus </=75 Years With Coronary Artery Disease Treated With COMBO Stents (From The MASCOT Registry). Am J Cardiol. 2020 Jul 15;127:1-8. doi: 10.1016/j.amjcard.2020.04.014. Epub 2020 Apr 24. PMID 32418717
- [Derived] Chandrasekhar J, Kerkmeijer LS, Kalkman DN, Sartori S, Aquino MB, Woudstra P, Beijk MA, Tijssen JG, Koch KT, Hajek P, Atzev B, Hudec M, Ong TK, Mates M, Borisov B, Warda HM, den Heijer P, Wojcik J, Iniguez A, Coufal Z, Khashaba A, Munawar M, Gerber RT, Yan BP, Lee M, Baber U, Dangas GD, Colombo A, de Winter RJ, Mehran R; MASCOT and REMEDEE investigators (full list of collaborators shown in the Appendix). Sex differences in 1-year clinical outcomes after percutaneous coronary intervention with COMBO stents: From the COMBO collaboration. Catheter Cardiovasc Interv. 2021 Apr 1;97(5):797-804. doi: 10.1002/ccd.28853. Epub 2020 Mar 21. PMID 32198837
- [Derived] Chandrasekhar J, Kalkman DN, Aquino MB, Sartori S, Hajek P, Atzev B, Hudec M, Ong TK, Mates M, Borisov B, Warda HM, den Heijer P, Wojcik J, Iniguez A, Coufal Z, Khashaba A, Schee A, Munawar M, Gerber RT, Yan BP, Tejedor P, Kala P, Liew HB, Lee M, Baber U, Vogel B, Dangas GD, Colombo A, de Winter RJ, Mehran R; MASCOT; REMEDEE investigators (Appendix I in the Supplementary material). 1-year results after PCI with the COMBO stent in all-comers in Asia versus Europe: Geographical insights from the COMBO collaboration. Int J Cardiol. 2020 May 15;307:17-23. doi: 10.1016/j.ijcard.2020.01.045. Epub 2020 Jan 24. PMID 32111358
- [Derived] Colombo A, Chandrasekhar J, Aquino M, Ong TK, Sartori S, Baber U, Lee M, Iniguez A, Hajek P, Borisov B, Atzev B, Den Heijer P, Coufal Z, Hudec M, Mates M, Snyder C, Moalem K, Morrell D, Elmore F, Rowland S, Mehran R; MASCOT Investigators. Safety and efficacy of the COMBO bio-engineered stent in an all-comer PCI cohort: 1-Year final clinical outcomes from the MASCOT post-marketing registry. Int J Cardiol. 2019 May 15;283:67-72. doi: 10.1016/j.ijcard.2019.01.053. Epub 2019 Jan 21. PMID 30826192